CLINICAL TRIAL: NCT02059616
Title: A Randomized, Double-blind, Multi-center, PhaseⅡ Clinical Trial to Evaluate the Antihypertensive Efficacy and Safety of Candesartan Cilexetil and Amlodipine Besylate for the Dose Selection in Patients With Essential Hypertension
Brief Title: A Phase 2 Dose Selection Trial of Candesartan Cilexetil and Amlodipine Besylate to Treat Essential Hypertension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_CCA_201
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Amlodipine; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- AML 5mg (Experimental): Amlodipine 5 mg, once a day for 8 weeks
  Interventions: Drug: Amlodipine 5mg
- AML 10mg (Experimental): Amlodipine 10 mg, once a day for 8 weeks
  Interventions: Drug: Amlodipine 10mg
- CC 8mg (Experimental): Candesartan Cilexetil 8 mg, once a day for 8 weeks
  Interventions: Drug: Candesartan Cilexetil 8mg
- CC 16mg (Experimental): Candesartan Cilexetil 16 mg, once a day for 8 weeks
  Interventions: Drug: Candesartan cilexetil 16mg
- AML 5mg/CC 8mg (Experimental): Amlodipine 5 mg and Candesartan 8 mg, once a day for 8 weeks
  Interventions: Drug: Amlodipine 5mg; Drug: Candesartan Cilexetil 8mg
- AML 5mg/CC16mg (Experimental): Amlodipine 5 mg and Candesartan Cilexetil 16 mg, once a day for 8 weeks
  Interventions: Drug: Amlodipine 5mg; Drug: Candesartan cilexetil 16mg
- AML 10mg/CC 8mg (Experimental): Amlodipine 10 mg and Candesartan Cilexetil 8 mg, once a day for 8 weeks
  Interventions: Drug: Amlodipine 10mg; Drug: Candesartan Cilexetil 8mg
- AML 10mg/CC 16mg (Experimental): Amlodipine 10 mg and Candesartan Cilexetil 16 mg, once a day for 8 weeks
  Interventions: Drug: Amlodipine 10mg; Drug: Candesartan cilexetil 16mg

INTERVENTIONS:
Drug: Amlodipine 5mg — Daily oral administration for 8 weeks
  Other Names: Norvasc 5mg
  Arms: AML 5mg; AML 5mg/CC 8mg; AML 5mg/CC16mg
Drug: Amlodipine 10mg — Daily oral administration for 8 weeks
  Other Names: Norvasc 10mg
  Arms: AML 10mg; AML 10mg/CC 16mg; AML 10mg/CC 8mg
Drug: Candesartan Cilexetil 8mg — Daily oral administration for 8 weeks
  Other Names: Atacand 8mg
  Arms: AML 10mg/CC 8mg; AML 5mg/CC 8mg; CC 8mg
Drug: Candesartan cilexetil 16mg — Daily oral administration for 8 weeks
  Other Names: Atacand 16mg
  Arms: AML 10mg/CC 16mg; AML 5mg/CC16mg; CC 16mg

SUMMARY:
The purpose of this study is to explore the optimal dose of fixed-dose combination of candesartan cilexetil and amlodipine besylate by examining the safety and efficacy of the combination therapy compared to each of the monotherapy in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 19 and ≤ 75 years old
* Subject with mild-to-moderate uncomplicated essential hypertension
* Subject who have voluntarily agreed to participate in the trial and signed the written informed consent form, after having listened to the purpose, method, and effect of the clinical trial

Exclusion Criteria:

* Subject with severe hypertension (siDBP ≥ 115 mmHg or siSBP ≥ 185 mmHg)
* Subject with difference in the mean blood pressure of over 10mmHg for siDBP or 20mmHg for siSBP between both arms at the screening visit
* Subject with known or suspected secondary hypertension [including but not limited to any of the following: renovascular hypertension, adrenal medullary and cortical hyperfunction, coarctation of the aorta, primary hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic kidney disease, etc.]
* Subject with symptomatic orthostatic hypotension (a sudden fall in siDBP of at least 10 mmHg or siSBP of at least 20 mmHg after standing compared with blood pressure from the sitting or supine position)
* Subject with Type 1 diabetes mellitus OR Type 2 diabetes mellitus with poor glucose control (defined as subject on insulin treatment, with HbA1c > 9.0%, or with a modification in the oral anti-hyperglycemic medication regiment within the past 12 weeks prior to Visit 1)
* Subject with severe heart disease (Congestive heart failure (NYHA Class III-IV), ischemic heart disease within the past 6 months (unstable angina, myocardial infarction), peripheral vascular disease, history of Percutaneous Transluminal Coronary Angioplasty or Coronary Artery Bypass Grafting)
* Subject with clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically significant arrhythmia
* Subject with hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, haemodynamically relevant stenosis of the aortic or mitral valve
* Subject with severe cerebrovascular disease (history of stroke, cerebral infarction, or cerebral hemorrhage within the past 6 months)
* Subject with or with a history of wasting disease, autoimmune diseases (rheumatoid arthritis, systemic lupus erythematosus), or connective tissue disease
* Subject with known moderate or malignant retinopathy (history of retinal signs of hemorrhage, visual impairment, retinal microaneurysm, etc. within the past 6 months)
* Subject with the following clinically significant laboratory abnormalities:

  * AST or ALT > 3 x Upper Limit Normal (ULN)
  * Serum Creatinine > 1.5 ULN
  * Serum potassium < 3.5 mmol/L or > 5.5 mmol/L
* Subject with any surgical or medical condition of the gastrointestinal tract that might significantly alter the absorption, distribution, metabolism or excretion of the drug
* Subject with a history of malignant tumors including leukemia and lymphoma within the past 5 years (except for localized basal cell carcinoma of the skin)
* Subject with any chronic inflammatory condition needing chronic anti-inflammatory therapy
* Subject with chronic kidney disease on dialysis
* Subject with cardiogenic shock
* Subject requiring concomitant use of other antihypertensive or contraindicated drugs during the entire study period
* Subject with known or suspected contraindications, including history of allergy or hypersensitivity to ARB or dihydropyridine derivatives
* Subject who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or ARB
* Pregnant women, lactating mothers, women suspected of being pregnant, women who wish to be pregnant during the study, or women of child-bearing potential who are not using medically acceptable methods of contraception (oral contraceptive, intra-uterine device, condom, etc.), except for women with surgical sterilization. Pre-menopausal women who are not surgically sterilized must have a negative pregnancy test result at Visit 1 and maintain acceptable methods of contraception throughout the study. Periodic abstinence (eg, symptothermal, calendar, post-ovulation methods), or hormonal contraceptive are not acceptable methods of contraception
* History of drug or alcohol abuse within the past 1 year
* Use of other investigational products within the past 4 weeks
* Subject who are judged unsuitable to participate in the study in the opinion of the investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in sitting Diastolic Blood Pressure (siDBP) at week 8 compared to baseline | Week 8

SECONDARY OUTCOMES:
Change in sitting Systolic Blood Pressure (siSBP) at week 4 and 8 | Week 4 and 8
Change in siDBP at week 4 | Week 4
Proportion of patients achieving ΔsiDBP > 10 mmHg and ΔsiSBP < 20 mmHg after 8 weeks | Week 8
Proportion of patients achieving siDBP < 90 mmHg and siSBP < 120 mmHg after 8 weeks | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jea Tahk, Principal Investigator — Ajou University School of Medicine
Locations (20):
- South Korea (20):
  - Seoul National University Bundang Hospital, Bundang
  - Dong-A University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Ilsan
  - Inha University Hospital, Incheon
  - Hallym University Sacred Heart hospital, Kyungki-do
  - Inje University Haeundae Baik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul Medical Center, Seoul
  - Seoul St. Mary's hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Yonsei University Gangnam Severance Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju